CLINICAL TRIAL: NCT04036253
Title: A Randomized, Comparative Study of HEMAX PFS® Versus EPREX/ ERYPO® in the Treatment of Anemia With Epoetin Alfa in Patients With Predialysis Chronic Kidney Disease
Brief Title: Study of HEMAX PFS Versus EPREX/ ERYPO® in Predialysis Chronic Kidney Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bio Sidus SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BIOS-HPFS-0115
Record Dates: First submitted 2019-07-12; First posted 2019-07-29 (Actual); Results first posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-02

CONDITIONS: Anemia of Chronic Kidney Disease
Keywords: epoetin; erythropoietin; Eprex; Hemax; Anemia; Chronic Kidney Disease; pre-dialysis
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eprex/Erypo (Active Comparator): Receive EPREX/ ERYPO® subcutaneously with an initial dose of 29 IU/ kg twice a week (2000 IU twice a week for 70 kg of weight), to be titrated according to the scheme that is summarized below.
  There will be a follow - up of patients with visits to the site every two weeks during the first 12 weeks of dose titration that will be followed by 12 additional weeks of dose maintenance with visits every 4 weeks.
  Interventions: Biological: Erythropoietin alfa
- Hemax PFS (Experimental): receive HEMAX® PFS subcutaneously with an initial dose of 29 IU/ kg twice a week (2000 IU twice a week for 70 kg of weight), to be titrated according to the scheme that is summarized below.
  There will be a follow - up of patients with visits to the site every two weeks during the first 12 weeks of dose titration that will be followed by 12 additional weeks of dose maintenance with visits every 4 weeks.
  Interventions: Biological: Erythropoietin alfa

INTERVENTIONS:
Biological: Erythropoietin alfa — Prefilled syringes of erythropoietin

SUMMARY:
Phase III, multicenter, randomized, open, controlled clinical trial. A study designed as phase III, in 120 patients with chronic renal failure in the pre-dialysis stage, evaluate efficacy and safety of Hemax PFS® (PFS: prefilled syringes) vs the innovator erythropoietin alfa product (Eprex®).

DETAILED DESCRIPTION:
This was a Phase IIIB, multicenter, randomized, open-label study to compare two products with epoetin alfa (HEMAX® PFS versus EPREX/ERYPO®).

This trial was open-label for both the patient and the investigator, but blinded in the performance of laboratory analyses.

The overall objective of the study was to evaluate the efficacy and the safety of HEMAX® PFS compared to EPREX/ERYPO®, following a dose-titration and maintenance scheme similar to the one used in the regular clinical practice.

All patients received HEMAX® PFS or EPREX/ERYPO® twice a week subcutaneously during 12 weeks of titration, switching then to an equivalent weekly dose during 12 additional maintenance weeks. During the dosing scheme switch from twice a week to once weekly, each patient continued receiving the treatment assigned at randomization.

The study conclude with n=43 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Patients with pre-dialysis chronic renal failure (CRF) defined by a glomerular filtration rate (calculated with the Modification of Diet in Renal Disease Study formula) ≥15 ml/ min and <60 ml/ min, by 1.73 m2
* Anemic patients that should be treated and levels of hemoglobin <10.5 g/dl and ≥ 7.5 g/dl.
* Patients that have the will and capacity to sign a written inform consent.
* Post-menopause women for at least 2 years, or sterile by surgery for at least 6 months. Women of childbearing age must have a negative pregnancy test at baseline and be willing to get an adequate method of contraception.

Exclusion Criteria:

* Patients that are planned to be on dialysis or have a renal transplant in the following 6 months.
* Transferrin iron Saturation < 20%.
* Etiology of renal failure (as secondary to autoimmune diseases) that, to the judge to the physician, can affect the normal development of the protocol.
* Active bleeding or history of hemorrhage that have led to a significative decrease of hematocrit in the last 30 days.
* Non-controlled hypertension (≥160 mm Hg of systolic pressure and/or ≥100 mm Hg of diastolic pressure with anti-hypertensive treatment).
* Anemia caused by any other cause than renal disease.
* Having a transfusion in the last 3 months before basal visit or during screening.
* Treatment with an erythropoiesis stimulant in the last 3 months before basal visit or screening.
* Increase risk of thromboembolic disease: history of arterial thromboembolia (stroke, transient ischemic attack, Acute coronary syndrome, etc.) in the last 6 months or venous in the last 12 months before screening; surgery in the last month before screening; prolong immobilization or orthopedic surgery programmed in the following 6 months or any other condition that to the judge of the investigator can increase the risk of thromboembolism.
* Hematological disease or myelodysplastic syndrome or history of hematological neoplasm or solid tumor in the last 5 years.
* History of congestive heart failure
* Pregnancy or breast feeding
* Refuse to participate in the protocol or any medical condition, that in the investigator opinion, is significant to prevent the participant from being included in the trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diego Ambrogetti, MD, Principal Investigator — Instituto de Investigaciones médicas Alfredo Lanari
Locations (11):
- Argentina (10):
  - CEMEDIC, Buenos Aires
  - CEREHA, Buenos Aires
  - CIMEL, Buenos Aires
  - CIPREC (Centro de Investigación y Prevención Cardiovascular), CABA
  - GEMA Consultorio, Caba
  - Hospital Argerich, CABA
  - Hospital Británico de Buenos Aires, CABA
  - Hospital Durand, CABA
  - Hospital Fernandez, CABA
  - Hospital Ramos Mejía, CABA
- IPHIC, Asunción, Paraguay

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Eprex/Erypo: Receive EPREX/ ERYPO® subcutaneously with an initial dose of 29 IU/ kg twice a week (2000 IU twice a week for 70 kg of weight), to be titrated according to the scheme that is summarized below.
  There will be a follow - up of patients with visits to the site every two weeks during the first 12 weeks of dose titration that will be followed by 12 additional weeks of dose maintenance with visits every 4 weeks.
  Erythropoietin alfa: Prefilled syringes of erythropoietin
- Hemax PFS: receive HEMAX® PFS subcutaneously with an initial dose of 29 IU/ kg twice a week (2000 IU twice a week for 70 kg of weight), to be titrated according to the scheme that is summarized below.
  There will be a follow - up of patients with visits to the site every two weeks during the first 12 weeks of dose titration that will be followed by 12 additional weeks of dose maintenance with visits every 4 weeks.
  Erythropoietin alfa: Prefilled syringes of erythropoietin
Period: Overall Study
Arm/Group | Eprex/Erypo | Hemax PFS
Started | 20 | 23
Completed | 16 | 20
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Eprex/Erypo | Hemax PFS | Total
Number analyzed (Participants) | 20 | 23 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 23 | 43
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 60.5 [20 to 80] | 64 [18 to 83] | 61 [18 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 17 | 32
  Male | 5 | 6 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 23 | 43
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Argentina | 17 | 22 | 39
  Paraguay | 3 | 1 | 4
Hemoglobin blood level [Mean (Standard Deviation); unit: g/dL] — Population: Three patients from the HEMAX group and four patients from the EPREX group did not complete the study procedures.
  g/dL
    number analyzed (Participants) | 18 | 22 | 40
    (all) | 9.56 (0.60) | 9.44 (0.81) | 9.50 (0.72)

OUTCOME MEASURES:

1. Primary Outcome: Efficacy Evaluation Through Change in Hemoglobin Levels
Description: Evaluate the efficacy of treatment with erythropoietin alfa through the measured changes in levels of hemoglobin from baseline value to the mean value of the 8 to 12 weeks of treatment, comparing patients treated with HEMAX® PFS versus EPREX/ ERYPO®.
Time Frame: 12 weeks of treatment
Population: Per protocol analysis
Measure: Mean (Standard Deviation); unit: Hemoglobin levels (g/dL)
Arm/Group | Eprex/Erypo | Hemax PFS
Number analyzed (Participants) | 20 | 23
Hemoglobin levels (g/dL)
  Baseline hemoglobin levels | 9.56 (0.60) | 9.44 (0.81)
  Average hemoglobin levels between visits 8 and 12 | 11.05 (0.74) | 11.11 (1.11)
  Hemoglobin levels change between both times | 1.49 (0.99) | 1.66 (1.05)

2. Primary Outcome: Adverse Events and Adverse Reactions (Safety and Tolerability) at Weeks 12 and 24.
Description: Evaluate the safety through the incidence of adverse events and adverse reactions asessed after 12 and 24 weeks of treatment (week 24 reported which includes those evaluated at week 12), comparing patients treated with HEMAX® PFS versus those treated with EPREX/ ERYPO®.
Time Frame: 24 weeks of treatment
Measure: Number; unit: Adverse Events
Arm/Group | Eprex/Erypo | Hemax PFS
Number analyzed (Participants) | 20 | 23
Adverse Events
  Overall Adverse Events | 23 | 30
  Serious Events | 4 | 4

3. Secondary Outcome: Percentage of Responder Patients
Description: Evaluate the efficacy of treatment with erythropoietin alfa through the percentage of responder patients (increase of Hb ≥ 1g/ dl) after 12 weeks of treatment, comparing patients treated with HEMAX® PFS versus those treated with EPREX/ ERYPO®.
Time Frame: 12 weeks of treatment
Population: Patients were classified as non-responders when hemoglobin did not increase at least 1 g/dL regarding baseline during any of the first 12 weeks of treatment
Measure: Number; unit: percentage of participants
Arm/Group | Eprex/Erypo | Hemax PFS
Number analyzed (Participants) | 18 | 22
percentage of participants
  Non-Responders | 5.56 | 4.55
  Responders | 94.44 | 95.45

4. Secondary Outcome: Percentage of Patients That Required Any Transfusion
Description: Evaluate the percentage of transfusional requirements after 12 weeks of treatment, comparing patients treated with HEMAX PFS versus those treated with EPREX/ ERYPO®.
Time Frame: 12 weeks of treatment
Measure: Number; unit: Percentage of patients
Arm/Group | Eprex/Erypo | Hemax PFS
Number analyzed (Participants) | 20 | 23
Percentage of patients | 5 | 0

5. Secondary Outcome: Change of Hemoglobin Level at Week 12 of Treatment
Description: Evaluate the efficacy between arms (HEMAX® PFS and EPREX/ ERYPO®) of treatment with erythropoietin alfa through the change in the level of hemoglobin from baseline in every visit until the week 12 visit.
Time Frame: Intragroup efficacy until week 12
Measure: Mean (Standard Deviation); unit: Hemoglobin levels (g/dL)
Arm/Group | Eprex/Erypo | Hemax PFS
Number analyzed (Participants) | 20 | 23
Hemoglobin levels (g/dL)
  Baseline | 9.56 (0.60) | 9.44 (0.81)
  Week 8 to 12 | 11.05 (0.74) | 11.11 (1.11)
  Change | 1.49 (0.99) | 1.66 (1.05)

6. Secondary Outcome: Evaluate the Efficacy Between Arms 24 Weeks: Week Doses in the Titration
Description: Evaluate the efficacy between arms (HEMAX® PFS and EPREX/ ERYPO®) of the change from the twice - a - week doses in the titration phase to a weekly dose in the maintenance phase through the changes in the hemoglobin levels from week 12 to weeks 16, 20 and 24 of treatment
Time Frame: Intragroup efficacy until week 24
Measure: Mean (Standard Deviation); unit: Hemoglobin levels (g/dL)
Arm/Group | Eprex/Erypo | Hemax PFS
Number analyzed (Participants) | 15 | 19
Hemoglobin levels (g/dL)
  Week 12 | 11.08 (0.9) | 11.16 (0.8)
  Week 16 | 10.9 (0.97) | 10.82 (1.12)
  Week 20 | 10.51 (0.90) | 10.71 (1.09)
  Week 24 | 10.97 (0.96) | 10.85 (1.44)

7. Secondary Outcome: Incidence of Anti-drug Antibodies (Immunogenicity)
Description: An anti-erythropoietin alfa antibody determination will be performed to evaluate treatment immunogenicity at week 12 and 24 visit
Time Frame: 12 and 24 weeks of treatment
Measure: Number; unit: Participants with positive result
Arm/Group | Eprex/Erypo | Hemax PFS
Number analyzed (Participants) | 20 | 23
Participants with positive result
  Week 12 | 0 | 0
  Week 24 | 0 | 1

8. Secondary Outcome: Concentration of Hepcidin
Description: Hepcidin will be analyzed by ELISA at baseline, week 12 and 24 in order to evaluate the treatment response.
Time Frame: 24 weeks of treatment
Population: The analysis was restricted to patients with available hepcidin samples at baseline, 12 weeks, and 24 weeks due to an unanticipated loss of samples.
Measure: Mean (Standard Deviation); unit: ng hepcidin/ml
Arm/Group | Eprex/Erypo | Hemax PFS
Number analyzed (Participants) | 10 | 14
ng hepcidin/ml
  Baseline | 84.80 (67.67) | 74.21 (64.26)
  Week 12 | 107.80 (96.31) | 56.07 (55.62)
  Week 24 | 83.60 (58.29) | 60.93 (44.16)

ADVERSE EVENTS:
Time Frame: After 12 and 24 weeks of treatment
Arm/Group | Eprex/Erypo | Hemax PFS
All-Cause Mortality (participants affected / at risk) | 1/20 | 0/23
Serious Adverse Events (participants affected / at risk) | 4/20 | 3/23
Other Adverse Events (participants affected / at risk) | 8/20 | 5/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eprex/Erypo (N=20) | Hemax PFS (N=23)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Worsening of renal function (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 2 (3)
Foot ulcer (Vascular disorders) | 0 (0) | 1 (1)
Worsened condition (General disorders) | 1 (1) | 0 (0) — Generalized implication syndrome, asthenia, frequent falls due to ambulatory difficulties, reason for which she was hospitalized.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eprex/Erypo (N=20) | Hemax PFS (N=23)
Increased blood pressure (Cardiac disorders) | 3 (3) | 3 (3)
Lower limb edema (Cardiac disorders) | 0 (0) | 2 (2)
Hypervolemia (Cardiac disorders) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0)
Acute diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Splenomegaly (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Increased lipids (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Increased creatinine levels (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Increased potassium levels (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Hypovitaminosis D (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Acute bronchitis (Infections and infestations) | 0 (0) | 2 (2)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Scabies (Infections and infestations) | 0 (0) | 1 (1)
Knee arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cervical pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Heel pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Insomnia (Nervous system disorders) | 1 (1) | 0 (0)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Increased body weight (General disorders) | 0 (0) | 1 (1)
Pruritus (General disorders) | 1 (1) | 0 (0)
Venous ulcer (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial disease (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-06-26): https://cdn.clinicaltrials.gov/large-docs/53/NCT04036253/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/53/NCT04036253/SAP_001.pdf